CLINICAL TRIAL: NCT03826875
Title: Preventative Treatment of Depression in Survivors of Aneurysmal Subarachnoid Hemorrhage
Brief Title: Poststroke Depression in Hemorrhagic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Michael Robert Levitt, MD, Assistant Professor, School of Medicine, Neurological Surgery, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00002718
Record Dates: First submitted 2019-01-28; First posted 2019-02-01 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Stroke Hemorrhagic; Depression
Keywords: stroke; hemorrhagic stroke; subarachnoid hemorrhage; depression
MeSH Terms: conditions — Hemorrhagic Stroke; Depression; Stroke; Subarachnoid Hemorrhage | interventions — Fluoxetine

STUDY DESIGN:
Intervention Model Description: double-blinded placebo-controlled randomized trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Patients randomized to the fluoxetine treatment group will be initially prescribed fluoxetine 20mg/day for a period of one year.
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator): Patients randomized to the placebo group will be initially prescribed placebo 20mg/day for a period of one year.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine — Patients who suffered aneurysmal subarachnoid hemorrhage will be prescribed fluoxetine and evaluated for the preventative treatment of depression and health-related quality-of-life
  Other Names: Prozac
  Arms: Treatment
Drug: Placebo — Patients who suffered aneurysmal subarachnoid hemorrhage will be prescribed placebo and evaluated for the preventative treatment of depression and health-related quality-of-life
  Arms: Placebo

SUMMARY:
A double-blinded placebo-controlled randomized trial to evaluate the effect of preventative treatment of depression in survivors of aneurysmal subarachnoid hemorrhage (aSAH), a type of stroke.

DETAILED DESCRIPTION:
Patients who suffered aneurysmal subarachnoid hemorrhage will be randomly assigned either an oral antidepressant or placebo and evaluated for the preventative treatment of depression and health-related quality-of-life.

ELIGIBILITY:
Inclusion Criteria:

Patients 18-85 years of age aged 18 years and older will be included.

Patients admitted for subarachnoid hemorrhage from a ruptured cerebral aneurysm will be included.

Only patients who provide informed consent will be included.

Exclusion Criteria:

Non-English speaking patients will be excluded.

Patients currently receiving therapy for depression or related mental health diagnoses before admission will be excluded.

Patients with medical contraindications to fluoxetine therapy will be excluded.

Pregnant patients or patients considering pregnancy during the trial period at the time of consent will be excluded.

Patients with active psychosis will be excluded.

Patients who are incarcerated or in police custody will be excluded.

Patients with a comorbidity or cognitive impairment (as determined by a recruiter-administered Montreal Cognitive Assessment; Patients scoring >26 are considered of appropriate cognitive function for consent) that precludes informed consent and participation in the research interviews will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levitt, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data provided.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo
- Drug Cohort: Fluoxetine 20mg/day
Period: Overall Study
Arm/Group | Placebo | Drug Cohort
Started | 4 | 4
Completed | 3 | 2
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Drug Cohort | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: year] | 50.75 (14.08) | 60.25 (9.74) | 55.50 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Baseline [Mean (Standard Deviation); unit: Score] — Population: HAM-D is a 21-item diagnostic/treating severe depression tool with only the first 17 items used (8 items scored 0-4, 9 scored 0-2; min-max: 0-50): 0-7 normal, 8-13 mild, 14-18 moderate, 19-22 severe, ≥23 very severe depression.
  PHQ-9 is a 9-item diagnostic/grading depression tool (min-max: 0-27): 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
  Score
    Hamilton Rating Scale for Depression (HAM-D) | 11.5 (10.61) | 8.67 (6.81) | 9.80 (7.33)
    Patient Health Questionnaire (PHQ-9) Depression | 10.25 (8.77) | 9.5 (6.81) | 9.88 (7.28)

OUTCOME MEASURES:

1. Primary Outcome: Depression
Description: Depression will be assessed using the Hamilton Rating Scale for Depression (HAM-D). The HAM-D is a 21-item questionnaire to treat and diagnose severe depression. Examining a different symptom or aspect of depression, such as mood, guilt feelings, or suicidal ideation. The first 17 questions are used for scoring. The first 17 items used (8 items scored 0-4, 9 scored 0-2; min-max: 0-50): 0-7 normal, 8-13 mild, 14-18 moderate, 19-22 severe, ≥23 very severe depression.
Time Frame: 1 year
Population: Patients withdrew
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Drug Cohort
Number analyzed (Participants) | 3 | 2
units on a scale | 12.33 (3.21) | 6 (5.66)

2. Primary Outcome: Depression
Description: Depression will be assessed using the Patient Health Questionnaire (PHQ-9). The PHQ-9 is a 9 item questionnaire to treat and diagnose depression. The minimum score is 1, and the maximum score is 27.
  1-4: minimal depression 5-9: mild depression 10-14: moderate depression 15-19: moderately severe depression 20-27: severe depression
Time Frame: 1 year
Population: patients withdrew
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Drug Cohort
Number analyzed (Participants) | 3 | 2
units on a scale | 5.67 (2.08) | 5.00 (7.07)

3. Secondary Outcome: Anxiety
Description: Anxiety will be assessed using the Hamilton Rating Scale for Anxiety. The Hamilton Anxiety Rating Scale measures the severity of anxiety through looking at both psychic and somatic anxiety. Each item is scored on a scale of 0 to 4, with a total range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Time Frame: 1 year
Population: patients withdrew
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Drug Cohort
Number analyzed (Participants) | 3 | 2
units on a scale | 8.00 (3.61) | 9.50 (6.36)

4. Secondary Outcome: Fatigue
Description: Fatigue will be assessed using the Fatigue Severity Scale. The Fatigue Severity Scale measures the severity of fatigue and its effect on a person's activities and lifestyle in patients exhibiting depression. The scale is designed to differentiate fatigue from clinical depression since they share similar symptoms. Scoring is done by calculating the average response to the question and people with depression typically score about 4.5 whereas those with fatigue average about 6.5.
  A minimum score is 1, and a maximum score is 7
  A score close to 4.5 is more likely to indicate depression. A score close to 6.5 is more likely to indicate fatigue.
Time Frame: 1 year
Population: patients withdrew
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Drug Cohort
Number analyzed (Participants) | 3 | 2
units on a scale | 2.71 (1.07) | 1.39 (0.08)

5. Secondary Outcome: Healthcare Utilization
Description: Healthcare Utilization will be assessed using the Self-Report Health Service Utilization and Medication Use. The Self-Report Health Service Utilization and Medication Use scale measures the frequency and purpose of healthcare utilization to include hospitalization, mental health care, inpatient admissions, outpatient visits, emergency room visits, skilled nursing facility/rehabilitation center visits, and medication usage. Scoring is the number of utilization per category per period.
  A minimum score is 0, and a maximum score is unlimited.
  A higher number indicates that the patient has utilized more health services and medication during 1 1-year time frame.
Time Frame: 1 year
Population: participants withdrew
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Drug Cohort
Number analyzed (Participants) | 3 | 2
units on a scale | 5.67 (8.46) | 23 (32.53)

6. Secondary Outcome: Social Support
Description: Social Support will be assessed using the Multidimensional Scale of Perceived Social Support (MSPSS). The MSPSS is a scale to determine a patient's social support system from Family, Friends, and significant other. The scale is comprised of a total of 12 items with 4 items for each subscale. The following subscale can also be calculated but not utilized in the report: Significant other average responses from questions 1,2,5,10; Family average responses from questions 3,4,8,11; friends average responses from questions 6,7,9,12.
  The total scale score is calculated by adding all 12 questions, then dividing by 12.
  A minimum score is 1, and a maximum score is 7.
  Total Scale Score of:
  1-2.9: low support 3-5: moderate support 5.1-7: high support
Time Frame: 1 year
Population: patients withdrew
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Drug Cohort
Number analyzed (Participants) | 3 | 2
units on a scale | 6.80 (0.34) | 4.75 (0.95)

7. Secondary Outcome: Sleep Disturbance
Description: (PROMIS-Sleep Disturbance). PROMIS is a sleep disturbance scale used to assess the pure domain of sleep disturbance. The short form is scored based on using a data collection tool that automatically calculates scores and will be using responses to each item for each participant. Scoring: The total raw score for a measure will be converted according to the PROMIS Score. The conversion table will translate the total raw score into a T-score for each participant. The T-score rescales the raw into a standardized score with a mean of 50 and a standard deviation of 10. Therefore, a person with a T-score of 40 is one standard deviation below the mean. A higher PROMIS T-score represents more of the concept being measured.
Time Frame: 1 year
Population: patients withdrew
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo | Drug Cohort
Number analyzed (Participants) | 3 | 2
T-score | 48.97 (9.35) | 44.85 (0.92)

8. Secondary Outcome: Function
Description: Function will be assessed using the The Short Form (18) Health Survey (SF-18). The SF-18is a 18-item questionnaire to assess health-related quality-of-life. Health concepts of physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Scoring: RAND scoring is composed of precoded numeric values that are recoded per RAND scoring key and each item is scored on a 0-100 range so that the lowest and highest possible scores are 0 and 100. Scores represent the percentage of total possible score achieved. In the second part of the scoring key, items are averaged together to create each scale allowing the scale to represent the average for all items in the scale that was answered.
Time Frame: 1 year
Population: patients withdrew
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Drug Cohort
Number analyzed (Participants) | 3 | 2
units on a scale | 78.40 (40.11) | 83.22 (10.65)

9. Secondary Outcome: Function
Description: Function will be assessed using the Barthel Index. The Barthel Index is a scale used to determine functional status, measuring performance in activities of daily living. Values assigned to each item are based on a time and amount of actual assistance required if a patient is unable to perform the activity. It can also be used to understand the course of rehabilitation and show how much progress toward independence has occurred. If there is a lack of improvement in the Barthel Index after a reasonable period of treatment, it indicates poor potential for rehab. The total score is not as significant or meaningful as the breakdown into individual items, but rather indicates where deficiencies are.
  A minimum score is 0, and a maximum score is 100.
  A patient scoring 0 is incontinent and cannot perform daily tasks independently.
  A patient scoring 100 is continent and able to perform daily tasks independently.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Drug Cohort
Number analyzed (Participants) | 3 | 2
units on a scale | 100 (0) | 100 (0)

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, an average of 1 year
Arm/Group | Placebo | Drug Cohort
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | Drug Cohort (N=4)
Meningitis (Surgical and medical procedures) | 1 (1) | 0 (0) — Repeat imaging showed no new bleeding. Symptoms of meningismus, headache, fever, and tachycardia, raising suspicion for meningitis and sepsis. Initially treated with 1L NS, antibiotics were switched from ceftriaxone to cefepime for broader coverage.

LIMITATIONS AND CAVEATS:
The number of participants enrolled was too low to draw a statistically significant result. Used 6-month follow-up data, as many participants did not complete the 12-month follow-up assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT03826875/Prot_SAP_000.pdf